CLINICAL TRIAL: NCT06872580
Title: A Phase I, Open-label, Dose Escalation and Expansion Study to Evaluate the Tolerability, Safety, Pharmacokinetics, and Initial Antitumor Activity of QLS1209 in Patients With Advanced Solid Tumors
Brief Title: A Study of QLS1209 in theTreatment of Patients With Advanced Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Qilu Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: QLS1209-101
Record Dates: First submitted 2025-03-05; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- QLS1209 mono dose escalation and optimization (Experimental)
  Interventions: Drug: QLS1209

INTERVENTIONS:
Drug: QLS1209 — Levels of QLS1209 will be explored in dose escalation, and determine the maximum tolerated dose.
Drug: QLS1209 — Every 21 days is one cycle.1-3 dose levels of QLS1209 will be explored in dose optimization, and determine the recommended dose (RD) of QLS1209 and evaluate the preliminary anti-tumor activity of QLS1209.

SUMMARY:
The goal of this clinical trial is to assess the safety and tolerability of QLS1209 alone in patients with eligible advanced solid tumors，determine the maximum tolerated dose (MTD) or maximum drug dose（MAD）of QLS1209, identify a recommended phase 2 dose (RP2D) and preferred schedule, examine preliminary pharmacokinetics (PK) and assess anti-tumor activity.

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in this clinical study; completely understand and know this study as well as sign the informed consent form (ICF);
* Age ≥ 18 years when ICF is signed;
* Eastern Cooperative Oncology Group performance status of 0 or 1;
* Expected survival ≥ 3 months;
* advanced malignant solid tumors who have failed standard treatment or have received no standard treatment；
* a) CCNE1 amplification determined by tumor or plasma next generation sequencing (NGS) or fluorescence in-situ hybridization (FISH); b) FBXW7 mutation determined by tumor or plasma NGS; c) PPP2R1A mutation determined by tumor or plasma NGS;
* Subjects with at least one evaluable tumor lesion (dose-escalation stage) or at least one measurable tumor lesion (dose-expansion stage) according to RECIST v1.1;

Exclusion Criteria:

* Previous treatment with PKMYT1 inhibitors;
* Received chemotherapy, biological therapy, endocrine therapy, immunotherapy, monoclonal antibody and other anti-tumor therapies within 4 weeks before the first dose of the investigational drug, special conditions are as follows:

  1. Including subjects who received oral fluorouracils, small molecule targeted drugs, radiotherapy or traditional Chinese medicines with anti-tumor indications within 2 weeks before the first dose;
  2. Including subjects who received treatment with mitomycin or nitrosoureas within 6 weeks before the first dose;
  3. Including subjects who received cell-based therapy or anti-tumor vaccines within 8 weeks before the first dose.
* Presence of uncontrolled or symptomatic central nervous system (CNS) metastases, or presence of leptomeningeal metastases or spinal cord compression due to metastases before signing the ICF. Exceptions: Subjects with symptomatic CNS metastases who have been treated and radiologically stable (defined as 2 brain images of the same imaging modalities, both acquired after treatment for brain metastases with an interval of at least 4 weeks, showing no intracranial progression by comparison) for ≥ 4 weeks before the first dose of the investigational drug, and have discontinued systemic sex hormone (any dose) therapy for > 2 weeks;
* Subjects with uncontrollable exudate or transudate (thoracic cavity, pericardium and abdominal cavity);
* Subjects with other active malignant tumors within 3 years before being included in the study (from the time of signing ICF), except for the following: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer, prostate cancer in situ, cervical cancer in situ, breast cancer in situ and other malignant tumors that have been treated without disease evidence within > 2 years and do not require continuous treatment; Known to be allergic to the investigational drug or any of its excipient;
* Subjects with current interstitial lung disease, pneumoconiosis, radiation pneumonitis, severely impaired lung function, etc. that may interfere with the monitoring and treatment of suspected drug-related pulmonary toxicity as judged by the investigator;
* Subjects who are unable to swallow and retain oral drugs, or have active gastrointestinal diseases (including inflammatory bowel disease and intestinal obstruction) and other conditions that seriously affect drug absorption as judged by the investigator;
* Subjects who have other serious physical or psychiatric diseases or laboratory test abnormalities that may increase the risk of participating in the study or interfere with the results of the study, and are considered unsuitable for participation in the study by the investigator;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
AEs, TEAEs, TRAEs, SAEs | up to 2 years
  Incidence, severity and relevance to the trial drug of adverse events (AEs), treatment-related adverse events (TEAEs), treatment-related adverse events (TRAEs) and serious adverse events (SAEs)
MTD/MAD | Up to 21 days after the first dose
  maximum tolerated dose/ maximum drug dose
RP2D | Up to 21 days after the first dose
  recommended phase II dose

SECONDARY OUTCOMES:
Tmax | up to 2 years
  Time to Reach Maximum (peak) Plasma Concentration Following Drug Administration
Cmax | up to 2 years
  Maximum Plasma Drug Concentration
ORR | up to 2 years
  Objective Response Rate
DoR | up to 2 years
  Duration of Response
DCR | up to 2 years
  Disease Control Rate
PFS | up to 2 years
  Progression-free Survival
OS | up to 2 years
  Overall Survival